CLINICAL TRIAL: NCT04790825
Title: Effect of Intensive or Conventional Periodontal Therapy on the Gut Microbiome and Systemic Inflammation of Patients With Inflammatory Bowel Disease: a Single-blinded Randomized Clinical Trial
Brief Title: Periodontal Therapy on the Gut Microbiome of Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBD-perio project
Record Dates: First submitted 2021-02-04; First posted 2021-03-10 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Periodontal Diseases; IBD; Dysbiosis; Inflammation
MeSH Terms: conditions — Periodontal Diseases; Dysbiosis; Inflammation | interventions — Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive periodontal treatment (Experimental): Adjunctive full-mouth intensive removal of subgingival dental plaque biofilms with the use of scaling and root planing after the administration of local anesthesia.
  Interventions: Procedure: Full mouth scaling and root planing (FMSRP)
- Community-based periodontal care (Active Comparator): Standard cycle of supragingival mechanical scaling and polishing.
  Interventions: Procedure: Full mouth scaling and root planing (FMSRP)

INTERVENTIONS:
Procedure: Full mouth scaling and root planing (FMSRP) — Subgingival instrumentation with ultrasonic devices and curettes of all periodontal pockets completed within 48 hours

SUMMARY:
Periodontitis and inflammatory bowel disease have been associated by meta-epidemiologic evidence, although their mechanistic connection needs to be further explored. Oral-gut axis is implicated in the pathogenesis of several chronic inflammatory conditions, but to date no studies have evaluated the impact of periodontal treatment on gut ecology. Thus, the present randomised clinical trial is aimed at investigating the effect of intensive or conventional periodontal therapy on the gut microbiome and parameters of systemic inflammation of patients diagnosed with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* clinical and instrumental diagnosis of ulcerative colitis or Crohn's disease
* periodontitis Stage III or IV
* BMI between 20 and 29 kg/m2
* free diet
* presence of at least 20 teeth

Exclusion Criteria:

* Systemic diseases (including diabetes, thyroid, liver, or kidney diseases)
* dietary allergies
* use of antibiotics or probiotics during the previous 30 days
* pregnancy or breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in microbiome alpha diversity measured from stool samples at 3 months | Baseline and 90 days
  Taxonomic and functional variation of gut bacteria after treatment

SECONDARY OUTCOMES:
Changes in microbiome alpha diversity measured from saliva samples at 3 months | Baseline and 90 days
  Taxonomic and functional variation of salivary bacteria after treatment
Change of the inflammatory markers levels in plasma | Baseline and 90 days
  Concentration of cytokines and biomarkers in plasma samples
Changes in mean clinical attachment level (CAL) at 3 months | Baseline and 90 days
  Variation in CAL after therapy assessed using a millimetre marked manual periodontal probe at 6 sites per tooth element
Changes in periodontal pocket depth (PPD) at 3 months | Baseline and 90 days
  Variation in PPD after therapy assessed using a millimetre marked manual periodontal probe at 6 sites per tooth element
Changes in full mouth bleeding score (FMBS) at 3 months | Baseline and 90 days
  Variation in the percentage of bleeding sites after therapy assessed by gentle probing at 6 sites per tooth element

CONTACTS AND LOCATIONS:
Locations (1):
- CIR Dental School, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided